CLINICAL TRIAL: NCT04105036
Title: Social Deprivation Assessment in Older Adults: Results From the Canadian Longitudinal Study on Aging
Brief Title: Social Deprivation Assessment in Older Adults
Status: Active, not recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, Principal Investigator, Jewish General Hospital
Other Study IDs: 2020-1956
Record Dates: First submitted 2019-09-23; First posted 2019-09-26 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Geriatrics; Social Deprivation
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- 45-54 years of age: Divided into two subgroups: individuals who are and are not socially deprived
  Interventions: Other: Data Collection
- 54-64 years of age: Divided into two subgroups: individuals who are and are not socially deprived
  Interventions: Other: Data Collection
- 65-74 years of age: Divided into two subgroups: individuals who are and are not socially deprived
  Interventions: Other: Data Collection
- 75-85 years of age: Divided into two subgroups: individuals who are and are not socially deprived
  Interventions: Other: Data Collection

INTERVENTIONS:
Other: Data Collection — Telephone interview questionnaire, in-home face-to-face interview, and data from the Collection Site

SUMMARY:
Social deprivation is a state to which older adults may be exposed, leading to adverse social, psychological, and health outcomes. Social deprivation may be more sensitive than socioeconomic status for predicting adversity while using only a few items for evaluation. However, there is no practical assessment for social deprivation in older Canadian adults. Two indices that capture a broad picture of social vulnerability have previously been developed for older Canadians. Using participants in the Canadian Longitudinal Study on Aging (CLSA), the overall objective is to examine and compare the associations of the COAD score and index, as well as the Keefe et al. and Andrew et al. indices with prevalent and incident adverse social, psychological, and health outcomes in participants at baseline assessment.

DETAILED DESCRIPTION:
Social deprivation is a state in which individuals are at risk for adverse health, as well as psychological and social outcomes. Social deprivation emphasises relative rather than absolute conditions, taking into account cultural standards of living in its classification of individuals. Increasing age is associated with increasing prevalence of social deprivation, putting older adults at risk for negative outcomes such as poor quality of life and ill-being. Rapid apprehension of social deprivation states by researchers and healthcare providers could improve management, favour proactivity, and increase understanding of health and social trends in older individuals.

No Canadian clinical assessment of social deprivation exists. There are only two social vulnerability indices that have been associated with incident health outcomes. On the other hand, the Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES: Évaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé) is a brief social deprivation assessment developed and validated in France. The Canadian Older Adult Deprivation (COAD) scale is a modified EPICES assessment. Using participants in the Canadian Longitudinal Study on Aging (CLSA), the global objective of this study is to examine whether the COAD score is in fact associated with social deprivation and its association with adverse social, psychological, and health outcomes.

Social deprivation is considered the state of an individual experiencing social withdrawal, poor economic conditions, and cultural deprivation; it exposes individuals to adverse social, health, and psychological outcomes. Social deprivation has been found to be influenced with many factors, including an individual's socioeconomic status (SES), gender, ethnicity and age, to name a few. The Canadian population is unique in its composition, with large immigrant, diverse, and ageing populations. This emphasises the need for a simple assessment specific to the Canadian population that can quickly yet accurately identify socially deprived older individuals. Currently, such a scale does not exist in the Canadian context. To bridge this gap, the French social deprivation assessment Evaluation of Deprivation and Inequalities in Health Examination Centres (EPICES: Évaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé) will be adapted to the Canadian context, creating the Canadian Older Adult Deprivation (COAD) scale. Moreover, as two Canadian social vulnerability and isolation indices have been previously created, the potential overlap between these indices and the COAD scale will be examined.

ELIGIBILITY:
Inclusion Criteria:

* Participants of the comprehensive CLSA assessment.

Exclusion Criteria:

* No information on social status
* No information on social, psychological, and health outcomes

Ages: 45 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals eligible for this study will be the participants of the CLSA
Sampling Method: Non-Probability Sample
Enrollment: 30000 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Social Deprivation | 1 day
  EPICES ( Évaluation de la Précarité et des Inégalités de santé dans les Centres d'Examens de Santé) scale, the cutoff 30.17 will be used

SECONDARY OUTCOMES:
Polypharmacy | 1 day
  The number of prescription medications taken on a daily basis, and in particular any number above 4 per day and the use of psychoactive drugs including benzodiazepines, antidepressants or neuroleptics
Comorbidities | 1 day
  Number of comorbidities
Mortality | 1 day
  Incident mortality
Depression | 1 day
  10 items from the Center for Epidemiological Studies' Short Depression Scale (CES-D) score ≥10
Falls | 1 day
  Number (if any) of falls
Mobility aid | 1 day
  Is a mobility aid used
Mobility | 1 day
  Difficulty walking 2 to 3 neighbourhood blocks
Activities daily living (ADL) | 1 day
  ADL score out of 6. Where a score of 3-5 is indicative of mild stages of neurocognitive disorders.
Instrumental activities of daily living (IADL) scales | 1 day
  IADL score out of 8. Where a score of 4-7 is indicative of mild stages of neurocognitive disorders.
Self-reported happiness, perception of health and mental health | 1 day
  Scored as excellent, very good, good, fair, or poor
Income | 1 day
  Personal income before tax
Social interaction/the availability of social support | 1 day
  Variables selected from the: social participation (SPA) questionnaire, social network (SN) questionnaire, social support availability (SSA) questionnaire
Place of living | 1 day
  Participants place of living is coded as home versus institution
Cognitive performance | 1 day
  Cognitive Module Assessment of the CLSA study from baseline assessment (e.g. the Animal Fluency Test)

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Undecided